CLINICAL TRIAL: NCT00139269
Title: Phase I/II Pilot Study of Induction Chemotherapy With Docetaxel in Combination With Cisplatin and 5-Fluorouracil (5-FU) in Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study of Docetaxel in Combination With Cisplatin and 5-Fluorouracil in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-199
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Advanced Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; SSCHN
Keywords: Advanced Squamous Cell Carcinoma; Squamous cell Carcinoma of Head and Neck; SSCHN; Docetaxel
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; Fluorouracil

INTERVENTIONS:
Drug: Docetaxel
Drug: Cisplatin
Drug: 5-Fluorouracil

SUMMARY:
The purpose of this study is to determine the appropriate dose, that dose which is found to give maximum effect with limited toxicity, of cisplatin in combination with docetaxel and 5-fluorouracil and then to further define the safety and effectiveness of this combination of medications.

DETAILED DESCRIPTION:
* Treatment begins with a one hour infusion of docetaxel followed by a 1/2 hour infusion of cisplatin. 5-fluorouracil will be administered through continuous IV infusion through a portable pump for four days at home. A cycle is twenty-one days long ( 4 days of chemotherapy and 17 days of recovery).
* During each cycle blood tests will be performed weekly. A physical exam will be performed and the impact of the chemotherapy will be assessed at the end of each cycle.
* If after 2 cycles the patients cancer has not responded sufficiently they will be removed from the study.
* If significant reduction in the size of the tumor is observed after cycle 2, a third and final cycle will be performed. Followed by radiation therapy twice daily for approximately 6-7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of head and neck (SSCHN).
* At least one bi- or uni-dimensionally measurable lesion.
* Stage II or IV disease without evidence of distant metastasis.
* No previous chemotherapy, radiotherapy or surgery (other than biopsy) for SSCHN.
* Age greater than 18 years.
* ECOG performance status of 0 or 1.
* Life expectancy of greater than 12 weeks.
* Adequate bone marrow, hepatic and renal function.
* Normal serum calcium

Exclusion Criteria:

* Primary tumor location in nasopharynx, nasal cavity, sinuses, or salivary glands.
* Patients with any non-SSCHN malignancy within 5 years of study entry, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix.
* Any prior treatment with chemotherapy.
* Prior radiotherapy to major bone marrow area (> 10% bone marrow) or to head and neck.
* Current peripheral neuropathy of greater than NCI grade 2.
* Other serious illness or medical condition
* Concurrent treatment with corticosteroids unless chronic treatment at low doses.
* Pregnant or lactating females or females of childbearing potential not employing adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 1998-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine whether cisplatin in combination with docetaxel and 5-fluorouracil can be given with acceptable side effects
to determine the efficacy of said combination.

SECONDARY OUTCOMES:
To define the safety profile, the dose limiting toxicity and the recommended dose of cisplatin in combination with docetaxel and 5-fluorouracil.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Principal Investigator — Dana-Farbar Cancer Institute

REFERENCES:
- [Background] Posner MR, Glisson B, Frenette G, Al-Sarraf M, Colevas AD, Norris CM, Seroskie JD, Shin DM, Olivares R, Garay CA. Multicenter phase I-II trial of docetaxel, cisplatin, and fluorouracil induction chemotherapy for patients with locally advanced squamous cell cancer of the head and neck. J Clin Oncol. 2001 Feb 15;19(4):1096-104. doi: 10.1200/JCO.2001.19.4.1096. PMID 11181674
- [Background] Haddad R, Colevas AD, Tishler R, Busse P, Goguen L, Sullivan C, Norris CM, Lake-Willcutt B, Case MA, Costello R, Posner M. Docetaxel, cisplatin, and 5-fluorouracil-based induction chemotherapy in patients with locally advanced squamous cell carcinoma of the head and neck: the Dana Farber Cancer Institute experience. Cancer. 2003 Jan 15;97(2):412-8. doi: 10.1002/cncr.11063. PMID 12518365